CLINICAL TRIAL: NCT03644667
Title: Targeting Inflammation and Alloimmunity in Heart Transplant Recipients With Tocilizumab (RTB-004)
Brief Title: Tocilizumab in Cardiac Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT RTB-004; ALL IN (Other: Study Team); U01AI136816 (NIH)
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Heart Transplant
Keywords: heart transplant recipients; alloimmunity; anti-inflammatory; tocilizumab; efficacy clinical trial; immunosuppression (IS)
MeSH Terms: interventions — tocilizumab; Calcineurin Inhibitors; Tacrolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab + Standard of Care Triple IS (Experimental): Tocilizumab plus standard of care triple immunosuppression (IS). Heart transplant recipients will receive tocilizumab (Actemra®) plus standard triple maintenance immunosuppression.
  Standard of care triple maintenance immunosuppression includes:
  * a calcineurin inhibitor (tacrolimus),
  * an anti-proliferative treatment (mycophenolate mofetil) or Myfortic® (enteric-coated mycophenolate sodium), and
  * steroids (methylprednisolone/prednisone) as prescribed by site physician investigator.
  Participants enrolled in the study will be followed for 24 months after their transplant surgery. Randomization will occur once a participant has weaned from cardiopulmonary bypass and has achieved hemodynamic stability without significant ongoing bleeding within the first 72 hours after transplant.
  Interventions: Biological: tocilizumab; Drug: Standard of Care Triple IS
- Placebo + Standard of Care Triple IS (Placebo Comparator): Placebo plus standard of care triple maintenance immunosuppression (IS). Heart transplant recipients will receive placebo plus standard triple maintenance immunosuppression.
  Standard of care triple maintenance immunosuppression includes:
  * a calcineurin inhibitor (tacrolimus),
  * an anti-proliferative treatment (mycophenolate mofetil) or Myfortic® (enteric-coated mycophenolate sodium), and
  * steroids (methylprednisolone/prednisone) as prescribed by site physician investigator.
  Participants enrolled in the study will be followed for 24 months after their transplant surgery. Randomization will occur once a participant has weaned from cardiopulmonary bypass and has achieved hemodynamic stability without significant ongoing bleeding within the first 72 hours after transplant.
  Interventions: Biological: Placebo; Drug: Standard of Care Triple IS

INTERVENTIONS:
Biological: tocilizumab — 6 doses: 8mg/kg (maximum of 800 mg) given once every four weeks by intravenous infusion over a 20-week period, with a minimum of 21 days between each infusion.
  Other Names: Actemra®
  Arms: Tocilizumab + Standard of Care Triple IS
Biological: Placebo — The placebo is 0.9% sterile normal saline. 6 doses: 8mg/kg (maximum of 800 mg) given once every four weeks by intravenous infusion over a 20-week period, with a minimum of 21 days between each infusion.
  Other Names: Placebo for tocilizumab; Placebo for Actemra®
  Arms: Placebo + Standard of Care Triple IS
Drug: Standard of Care Triple IS — Standard of care triple maintenance IS includes:
  1. A calcineurin inhibitor-tacrolimus (Prograf ®) per site standards by sublingual, oral or intravenous route to attain target trough levels.
     Exception: Should a participant be unable to tolerate tacrolimus, the site physician investigator may choose cyclosporine treatment.
  2. An anti-proliferative treatment-mycophenolate mofetil or Myfortic® (enteric-coated mycophenolate sodium) will be administered, per protocol.
     Exception: Should a participant be unable to tolerate mycophenolate mofetil, the site physician investigator may choose an alternative treatment.
  3. Steroids-methylprednisolone/prednisone dosing will be given according to the local center standard of practice early post transplantation. After 6 months, prednisone may be withdrawn at the discretion of the site physician investigator, per protocol.
  Other Names: calcineurin inhibitor: (tacrolimus (Prograf ®)); anti-proliferative treatment: (mycophenolate mofetil ),; MMF, CellCept®; Myfortic®, enteric-coated mycophenolate sodium; steroids: methylprednisolone/prednisone

SUMMARY:
The purpose of this research study is to see if a study drug called Tocilizumab will, when given with standard anti-rejection medicines, lead to better heart transplantation outcomes at 1 year after the transplant. Specifically, the investigators will evaluate whether taking tocilizumab leads to less rejection, less development of unwanted antibodies, and better heart function.

DETAILED DESCRIPTION:
This is a prospective, multi-center phase 2 clinical trial in which 200 primary heart transplant recipients will be randomized (1:1) to receive either tocilizumab (Actemra®) or placebo (normal saline) plus standard triple maintenance immunosuppression. Investigators will recruit primary heart transplant recipients from 14 participating centers. Subjects will be screened, consented, and enrolled while on the United Network for Organ Sharing (UNOS) wait list. When the recipient has received the transplant and is deemed hemodynamically stable, randomization will occur.

Study duration: The study duration will be approximately 4 years. There will be a 36-month accrual period, and participants will be followed for a minimum 12-month, and a maximum 24 months after heart transplantation.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases does not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria- Study Entry

1. Subject must be able to understand and provide informed consent;
2. Is a candidate for a primary heart transplant (listed as a heart transplant only);
3. No desensitization therapy prior to transplant;
4. Agreement to use contraception: according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective.

   * Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from the above referenced list to be used for the duration of the study
   * Those who choose oral contraception must agree to use a second form of contraception after administration of study drug for a period of 1 year after the last dose of study drug.
5. Mechanical support or investigational drug trials where the intervention ends at the time of transplantation are permitted;
6. In the absence of contraindication, vaccinations should be up to date for hepatitis B, influenza, pneumococcal, zoster, and Measles, Mumps, & Rubella (MMR); and
7. Subjects from areas of endemic coccidioidomycosis are eligible for inclusion but must be treated prophylactically with fluconazole or itraconazole.

Inclusion Criteria - Randomization

1. Recipient of a primary heart transplant;
2. Negative virtual crossmatch (according to local center criteria);
3. No desensitization therapy prior to transplant;
4. Female subjects of childbearing potential must have a negative pregnancy test (serum or urine) prior to randomization; and
5. Agreement to use contraception: according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective.

   * Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from the above referenced list to be used for the duration of the study
   * Those who choose oral contraception must agree to use a second form of contraception after administration of study drug for a period of 1 year after the last dose of study drug.
6. Negative SARS-CoV-2 real-time reverse transcription polymerase chain reaction (rRT-PCR) test result performed within 48 hours of transplant (SARS-CoV-2 is the virus that causes COVID-19)

Exclusion Criteria:

Exclusion Criteria Study Entry

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
2. Candidate for a multiple solid organ or tissue transplants;
3. Prior history of organ or cellular transplantation requiring ongoing systemic immunosuppression;
4. Currently breast-feeding a child or plans to become pregnant during the timeframe of the study follow up period;
5. History of severe allergic and/or anaphylactic reactions to humanized or murine monoclonal antibodies;
6. Known hypersensitivity to tocilizumab (Actemra®);
7. Previous treatment with tocilizumab (Actemra®);
8. Human Immunodeficiency Virus (HIV) positive;
9. Hepatitis B surface antigen positive;
10. Hepatitis B core antibody positive;
11. Hepatitis C virus antibody positive (anti-HCV Ab+) who are either untreated or, have failed to demonstrate sustained viral remission for more than 12 months (after anti-viral treatment);
12. Recipient of a Hepatitis C virus nucleic acid test (NAT) positive donor organ;
13. Subjects must be tested for latent TB infection (LTBI) within a year prior to transplant:

    --Subjects with a positive test for LTBI must complete appropriate therapy for LTBI.

    ---A Subject is considered eligible only if they have a negative test for LTBI within one year prior to transplant OR

    ---- if they have completed appropriate LTBI therapy within one year prior to transplant.
14. Subjects with a previous history of active Tuberculosis (TB);
15. Subjects with a history of splenectomy;
16. Known active current viral, fungal, mycobacterial or other infections not including (left ventricular assist device [LVAD]) driveline infections;
17. History of malignancy less than 5 years in remission.

    --Any history of adequately treated in-situ cervical carcinoma, low grade prostate carcinoma, or adequately treated basal or squamous cell carcinoma of the skin will be permitted.
18. History of hemolytic-uremic syndrome/ thrombotic thrombocytopenia purpura;
19. History of demyelinating disorders such as:

    * multiple sclerosis,
    * chronic inflammation,
    * demyelinating polyneuropathy.
20. History of gastrointestinal perforations, active inflammatory bowel disease or diverticulitis;
21. Any previous treatment with alkylating agents such as chlorambucil or, total lymphoid irradiation;
22. Radiation therapy within 3 weeks before enrollment.

    --Enrollment of subjects who require concurrent radiotherapy should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
23. Subjects with a hemoglobin <7.0gm/dL (last measurement within 7 days prior to transplant);
24. Subjects with a platelet count of less than 100,000/mm^3 (last measurement within 7 days prior to transplant);
25. Subjects with an absolute neutrophil count (ANC) of less than 2,000/mm^3 (last measurement within 7 days prior to transplant);
26. Subjects with Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) levels >3 x Upper Limit of Normal (ULN);
27. Subjects who are administered or intended to be administered cytolytic or anti-cluster of differentiation 25 (CD25) monoclonal antibody agents as induction therapy in the immediate post-transplant period;
28. Intent to give the recipient a live vaccine within 30 days prior to randomization;
29. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may:

    * pose additional risks from participation in the study,
    * may interfere with the participant's ability to comply with study requirements, or
    * that may impact the quality or interpretation of the data obtained from the study.

Exclusion Criteria - Randomization

1. Recipient of multiple solid organ or tissue transplants;
2. Recipient of ex vivo preserved hearts and hearts donated after cardiac death (DCD);
3. Currently breast-feeding a child or plans to become pregnant during the timeframe of the study follow up period;
4. History of severe allergic anaphylactic reactions to humanized or murine monoclonal antibodies;
5. Known hypersensitivity to tocilizumab (Actemra®);
6. Previous treatment with tocilizumab (Actemra®);
7. HIV positive;
8. Hepatitis B surface antigen positive;
9. Hepatitis B core antibody positive;
10. Hepatitis B negative transplant recipient that received a transplant from a hepatitis B core antibody positive donor;
11. HCV+ subject(s) who are either untreated or have failed to demonstrate sustained viral remission for more than 12 months after anti-viral treatment;
12. Recipient of a hepatitis C virus nucleic acid test (NAT) positive donor organ;
13. Subject's organ donor tests positive for SARS-CoV-2 by real-time reverse transcription polymerase chain reaction (SARS-CoV-2 is the virus that causes COVID-19).
14. Subjects with a previous history of active (TB);
15. Subjects must be tested for latent TB infection (LTBI) within a year prior to transplant:

    --Subjects with a positive test for LTBI must complete appropriate therapy for LTBI.

    ---A Subject is considered eligible only if they have a negative test for LTBI within one year prior to transplant OR

    ---- if they have completed appropriate LTBI therapy within one year prior to transplant.
16. Subjects with a history of splenectomy;
17. Known active current viral, fungal, mycobacterial or other infections, not including (left ventricular assist device [LVAD]) driveline infections;
18. History of malignancy less than 5 years in remission.

    --Any history of adequately treated in-situ cervical carcinoma, low grade prostate carcinoma, or adequately treated basal or squamous cell carcinoma of the skin will be permitted.
19. History of hemolytic-uremic syndrome/ thrombotic thrombocytopenia purpura;
20. History of demyelinating disorders;
21. History of gastrointestinal perforations, active inflammatory bowel disease or diverticulitis;
22. Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation;
23. Radiation therapy within 3 weeks before randomization.

    --Enrollment of subjects who require concurrent radiotherapy should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
24. Subjects with a hemoglobin <7.0gm/dL within 7 days prior to randomization;
25. Subjects with a platelet count of less than 100,000/mm^3 within 7 days prior to randomization;
26. Subjects with an absolute neutrophil count (ANC) of less than 2,000/mm^3 within 7 days prior to randomization;
27. Subjects with AST or ALT levels >3 x ULN;
28. Subjects who are administered or intended to be administered cytolytic or anti- CD25 monoclonal antibody agents as induction therapy in the immediate post- transplant period;
29. Receipt of a live vaccine within 30 days prior to randomization;
30. Use of investigational drugs after transplantation;
31. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator,

    * may pose additional risks from participation in the study,
    * may interfere with the participant's ability to comply with study requirements, or
    * that may impact the quality or interpretation of the data obtained from the study.
32. Subjects with known donor-specific antibody at the time of evaluation of antibodies for heart transplant surgery (within 6 months).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Positive for Event of dnDSA, ACR, AMR, Hemodynamic Compromise, Death or Re-Transplantation - By Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  This outcome is defined by a composite 1 year post-transplant endpoint of:
  * detection of de novo donor-specific antibodies (dnDSA) (Core Laboratory),
  * acute cellular rejection (ACR) ≥ ISHLT 2R rejection (Core Laboratory),
  * antibody mediated rejection (AMR) ≥ ISHLT AMR 1 (Core Laboratory),
  * hemodynamic compromise rejection in the absence of a biopsy or histological rejection,
  * death, or
  * re-transplantation.

SECONDARY OUTCOMES:
Freedom of Detection of de Novo Donor-Specific Antibodies (dnDSA) - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  A comparison by treatment group of the incidence of freedom from development of de novo donor-specific antibodies (dnDSA). dnDSA is a newly developed alloantibody that is against the donor organ.
Freedom from Acute Cellular Rejection (ACR) ≥ International Society of Heart and Lung Transplantation (ISHLT) 2R Rejection - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  A comparison by treatment group of the incidence of freedom from development of acute cellular rejection ≥2R (Reference: International Society of Heart and Lung Transplantation [ISHLT] acute cellular rejection-grade 2R or greater severity).
Freedom from Antibody Mediated Rejection (AMR) ≥ International Society of Heart and Lung Transplantation (ISHLT) AMR 1 - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  A comparison by treatment group of the incidence of freedom from development of antibody-mediated rejection defined as ISHLT grade AMR 1 or greater severity.
Freedom from Hemodynamic Compromise Rejection in the Absence of a Biopsy or Histological Rejection - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  A comparison by treatment group of the incidence of freedom from development of hemodynamic compromise (HDC).
  Hemodynamic compromise is defined by:
  - Need for inotropic agents due to a Cardiac Index (CI) <2.0 L/min/m^2 or a 25% decrease from baseline, in addition to one of the following:
  * ejection fraction of <40% or a 20% decrease from baseline, and the need for inotropic agents OR
  * fractional shortening of <20% or a 25% decrease from baseline, and the need for inotropic agents.
Freedom from Any-Treated Rejection - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  A comparison by treatment group of the incidence of freedom from development of episode of rejection requiring treatment. Reference: Acute cellular rejection as defined by the 2004 International Society of Heart and Lung Transplantation (ISHLT) grading scale.
Freedom from Acute Cellular Rejection (ACR) ≥ International Society of Heart and Lung Transplantation (ISHLT) 2R Per Patient - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  A comparison by treatment group of the incidence of freedom from acute cellular rejection (ACR) ≥ ISHLT 2R rejection. Reference: 2004 International Society of Heart and Lung Transplantation [ISHLT [ grading scale).
Freedom from Antibody Mediated Rejection (AMR) (≥ International Society of Heart and Lung Transplantation (ISHLT) AMR 1) Per Participant - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)]
  Time from transplant, free of antibody mediated rejection, defined as ISHLT grade AMR 1 or greater will be compared between the treatment groups. Hemodynamic compromise is defined as the need for inotropic agents due to a Cardiac Index (CI) <2.0 L/min/m2 or a 25% decrease from baseline in addition to one of the following:
  * Ejection fraction of <40% or a 20% decrease from baseline, and the need for inotropic agents
  * Fractional shortening of <20% or a 25% decrease from baseline, and the need for inotropic agents
Freedom from Hemodynamic Compromise Rejection in the Absence of a Biopsy or Histological Rejection Per Participant - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  Time from transplant, free of antibody mediated rejection, defined as ISHLT grade AMR 1 or greater will be compared between the treatment groups
Occurrence of Death - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  Incidence of all-cause mortality will be compared between the treatment groups.
Occurrence of Re-Listed for Transplantation - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)
  Incidence of participant(s) being re-listed for transplant will be compared between the treatment groups.
Occurrence of Re-Transplantation - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)]
  Incidence of participant(s) re-transplantation will be compared between the treatment groups.
Number of Acute Cellular Rejection (≥ International Society of Heart and Lung Transplantation (ISHLT) 2R) Per Patient - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)]
  The frequency of events will be compared between the treatment groups.
Number of Antibody Mediated Rejection (AMR) (≥ International Society of Heart and Lung Transplantation (ISHLT) AMR 1) Per Participant - by Treatment Group | 12 months post-transplantation
  The frequency of events will be compared between the treatment groups.
Number of Rejection Episodes Associated with Hemodynamic Compromise (HDC) Per Participant - by Treatment Group | From transplant through 12 months post transplant surgery (12 months)]
  The frequency of events will be compared between the treatment groups.
Change in Intravascular Ultrasound (IVUS) Measurements From Baseline to 1 Year Post-Transplant- by Treatment Group | Baseline (4 to 8 weeks post-transplant), 1 year post-transplant
  Per protocol, per clinical research site standard of care.
Angiographic Evidence of Cardiac Allograft Vasculopathy (CAV) - by Treatment Group | 12 months post-transplantation
  In accordance with the International Society of Heart and Lung Transplantation (ISHLT) Cardiac Allograft Vasculopathy (CAV) angiographic grading scale.
Participant Loss to follow up - by Treatment Group | 12 months post-transplantation
  Incidence of participant loss to follow up will be compared between the treatment groups.
Occurrence of Serious Infections Requiring Intravenous Antimicrobial Therapy and Need for Hospitalization - by Treatment Group | Through 24 months post transplant surgery
  The frequency of serious infections requiring intravenous antimicrobial therapy and need for hospitalization will be compared between treatment groups.
Incidence of Tuberculosis - by Treatment Group | Through 24 months post transplant surgery
  The incidence of tuberculosis will be compared between treatment groups.
Incidence of Cytomegalovirus (CMV) Infection - by Treatment Group | Through 24 months post transplant surgery
  The incidence of CMV infection will be compared between treatment groups.
Incidence of Post-Transplant Lymphoproliferative Disease (PTLD) - by Treatment Group | Through 24 months post transplant surgery
  The incidence of PTLD will be compared between treatment groups.
Tolerability (Discontinuation of Study Drug) of Tocilizumab (TCZ) - by Treatment Group | Through 24 months post transplant surgery
  The number of participants who discontinue study drug, per protocol, will be compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jon A. Kobashigawa, MD, Study Chair — Cedars Sinai Medical Center: Transplantation; Joren C. Madsen, MD, DPHIL, Principal Investigator — Massachusetts General Hospital: Transplantation
Locations (20):
- United States (20):
  - Cedars Sinai Medical Center (CACS), Beverly Hills, California
  - University of California, San Diego: Sulpizio Cardiovascular Center (CASD), La Jolla, California
  - Stanford Health Care (CASU), Stanford, California
  - Tampa General Hospital (FLTG), Tampa, Florida
  - Northwestern Memorial Hospital (INLM), Chicago, Illinois
  - Tufts Medical Center (MANM), Boston, Massachusetts
  - Massachusetts General Hospital (MAMG), Boston, Massachusetts
  - St. Luke's Hospital of Kansas City (MOLH), Kansas City, Missouri
  - University of Nebraska Medical Center (NEUN), Omaha, Nebraska
  - Mount Sinai Medical Center (NYMS), New York, New York
  - Columbia University Medical Center (NYCP), New York, New York
  - Montefiore Medical Center (NYMA), The Bronx, New York
  - Duke University Medical Center (NCDU), Durham, North Carolina
  - Cleveland Clinic Foundation (OHCC), Cleveland, Ohio
  - Penn State Health: Milton S. Hershey Medical Center (PAHE), Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania (PAUP), Philadelphia, Pennsylvania
  - Allegheny General Hospital (PAAG), Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center (TNVU), Nashville, Tennessee
  - Baylor University Medical Center (TXTX), Dallas, Texas
  - University of Utah (UTMC), Salt Lake City, Utah

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: The Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait